CLINICAL TRIAL: NCT02194023
Title: Inhibition of de Novo Plaque Formation and Side Effects of Two New Mouthrinse Formulations: 0.12% and 0.03% Chlorhexidine Digluconate, Respectively, in a 4-day Non-brushing Model. A Triple-blind, Randomized Clinical Trial.
Brief Title: Clinical Effects of Two New Chlorhexidine Digluconate Formulations: 0.12% and 0.03%.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Dentaid SL (Industry)
Responsible Party: Principal Investigator, Carolina Mor, Master in periodontics by Universitat Internacional de Catalunya., Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PER-ECL-2011-06-NF
Record Dates: First submitted 2014-07-13; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Dental Plaque; Side Effects
Keywords: chlorhexidine digluconate; gingivitis; cetylpyridinium chloride; mouthrinse; dental plaque; de novo; in vivo
MeSH Terms: conditions — Dental Plaque; Gingivitis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (PCB) (Placebo Comparator): Placebo mouthrinse: physiological saline solution (0.9% w/w solution of NaCl in deionized water)
  Interventions: Drug: Placebo: PCB
- 0.12%NF (Experimental): 0.12% Chlorhexidine digluconate new formulation
  Interventions: Drug: 0.12%NF
- 0.03%NF (Experimental): 0.03% Chlorhexidine digluconate new formulation
  Interventions: Drug: 0.03%NF
- PAT (Perio-Aid Treatment) (Active Comparator): Commercialized 0.12% Clorhexidine digluconate (Perio-Aid Treatment, Dentaid, Spain)
  Interventions: Drug: PAT

INTERVENTIONS:
Drug: Placebo: PCB — Participants were asked to rinse every 12 hours, with 15 ml for 30 seconds, and after spitting to refrain from rinsing their mouths with water and from eating or drinking for at least 60 minutes.
  Other Names: saline solution
  Arms: Placebo (PCB)
Drug: 0.12%NF — Participants were asked to rinse every 12 hours, with 15 ml for 30 seconds, and after spitting to refrain from rinsing their mouths with water and from eating or drinking for at least 60 minutes.
  Arms: 0.12%NF
Drug: 0.03%NF — Participants were asked to rinse every 12 hours, with 15 ml for 30 seconds, and after spitting to refrain from rinsing their mouths with water and from eating or drinking for at least 60 minutes.
  Arms: 0.03%NF
Drug: PAT — Patients were asked to rinse every 12 hours, and after spitting to refrain from rinsing their mouths with water and from eating or drinking for at least 60 minutes.
  Other Names: Perio-Aid Treatment
  Arms: PAT (Perio-Aid Treatment)

SUMMARY:
In the current study we tested the hypothesis that new 0.05% Cetylpyridinium chloride (CPC) mouthrinse formulations containing 0.12% or 0.03% chlorhexidine digluconate (CHX): 1) yield similar or better clinical results regarding the inhibition of de novo plaque growth compared to those achieved with an already marketed 0.12% CHX mouthrinse (Perio-Aid Treatment without alcohol. Dentaid, Spain), 2) reduce the side effects caused by the marketed 0.12% CHX formula and 3) that these mouthrinses have no negative microbiological effects, and they control total bacterial loads.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years
* Good overall health without medical history or medications that could interfere with the study conduct.
* Minimum of 6 teeth per quadrant.
* Absence of probing depths ≥4mm.

Exclusion Criteria:

* Allergy to CHX or to CPC.
* Continuous use of CHX or of any other oral antiseptic in the months prior to the study.
* Any adverse medical background or long-term medications that could affect gingival conditions.
* Having taken antibiotics in the previous three months.
* Moderate to severe gingivitis (bleeding on probing ≥ 40%). 41(Van der Weijden et al. 1994).
* Pregnancy or breastfeeding.
* Smokers of more than 5 cigarettes per day.
* Orthodontic appliances.
* Fixed or removable prostheses.
* Systemic diseases that increase the risk for gingival diseases (diabetes mellitus, immunosuppression).
* Severe dental crowding.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with greater reduction of plaque regrowth and side effects. | Baseline to 4 days.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Mor-Reinoso, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- UIC dental office, Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona, Spain